CLINICAL TRIAL: NCT06872697
Title: The Effect of Whole Body Vibration Application on Muscle Functional Level and Respiratory Parameters in Intensive Care Patients
Brief Title: Impact of Whole Body Vibration on Muscle Function and Respiratory Parameters in Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Elif Kabasakal, LECTURER, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4/2023.K-11
Record Dates: First submitted 2024-12-20; First posted 2025-03-12 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Intensive Care Patients; Whole Body Vibration
MeSH Terms: interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- whole body vibration group (Experimental): In the group receiving whole-body vibration in addition to conventional treatment, the whole-body vibration will be performed with the patient's hips and knees in approximately 20° flexion, and the bed inclined to 25-30°. The vibration platform will be fixed at the end of the bed, and the patients will apply pressure with their feet on the platform. The whole-body vibration will be administered for 3 minutes, 1-4 sets, at a frequency of 20-25 Hz, 5 days a week, for 4 weeks.
  Interventions: Other: whole body vibration; Other: Conventional Physiotherapy
- Neuromuscular Electrical Stimulation Group (Active Comparator): In addition to conventional treatment, low-frequency neuromuscular electrical stimulation with a symmetrical biphasic waveform at 50 Hz will be applied to the biceps brachii and quadriceps femoris muscles for 45 minutes per session, 5 days a week, for 4 weeks.
  Interventions: Device: Neuromuscular Electrical Stimulation; Other: Conventional Physiotherapy
- control group (Active Comparator): As conventional treatment (CT), normal range of motion exercises, airway clearance techniques, breathing exercises, and mobilization will be applied 5 days a week for 4 weeks.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: whole body vibration — In the group receiving whole-body vibration in addition to conventional treatment, the whole-body vibration will be performed with the patient's hips and knees in approximately 20° flexion, and the bed inclined to 25-30°. The vibration platform will be fixed at the end of the bed, and the patients will apply pressure with their feet on the platform. The whole-body vibration will be administered for 3 minutes, 1-4 sets, at a frequency of 20-25 Hz, 5 days a week, for 4 weeks, depending on the protocol, in addition to conventional physiotherapy.
  Arms: whole body vibration group
Device: Neuromuscular Electrical Stimulation — In this group, neuromuscular electrical stimulation (NMES) will be applied to the targeted muscle groups. The application will be carried out with the patient in a comfortable seated or lying position. Stimulation parameters will be set as follows: a frequency of 35-50 Hz, a pulse duration of 200-400 microseconds, and an intensity adjusted to elicit visible muscle contractions without causing discomfort. NMES will be applied for 20-30 minutes per session, 3-5 times a week, for 4-6 weeks, depending on the protocol, in addition to conventional physiotherapy.
  Other Names: electrotherapy
  Arms: Neuromuscular Electrical Stimulation Group
Other: Conventional Physiotherapy — The conventional treatment program will include normal range of motion, airway clearance techniques, breathing exercises, and mobilization.

SUMMARY:
Immobility and mechanical ventilation in intensive care unit (ICU) patients lead to muscle weakness and loss, particularly in antigravity and respiratory muscles. Early physiotherapy interventions are crucial to prevent complications, reduce side effects, shorten intubation time, and lower patient costs. ICU physiotherapy includes chest physiotherapy, range of motion exercises, strengthening exercises, mobilization, positioning, and inspiratory/peripheral muscle training.

Muscle training plays a key role in ICU physiotherapy. Whole Body Vibration (WBV) is a promising, side-effect-free intervention to enhance muscle strength in various populations. Its effects result from neuromuscular responses to mechanical vibrations and the tonic vibration reflex. WBV has been reported to improve muscle strength, elasticity, circulation, and balance while reducing pain and fall risk. However, its effects on ICU patients remain unclear. To date, only one study has shown increased muscle electrical activity in ICU patients after WBV, but no research has evaluated changes in muscle strength, mass, or elasticity.

Another method used in muscle training is neuromuscular electrical stimulation (NMES), which prevents muscle atrophy, strengthens muscles, and restores endurance. NMES is suitable for patients with limited cooperation, making it an alternative to active exercise. No study has compared NMES and WBV in immobile ICU patients. Given the limited non-pharmacological options in ICU care, particularly for unconscious or uncooperative patients, identifying effective alternatives is essential.

This study aims to compare the effects of WBV and NMES on respiratory muscle strength, respiratory parameters, and muscle mass, composition, elasticity, and strength in ICU patients. Participants will be divided into three groups: WBV (n=15), NMES (n=15), and conventional therapy only (n=15). All groups will receive conventional therapy five days a week for four weeks, with WBV added to the first group and NMES to the second. Functional status, muscle assessments, grip strength, respiratory muscle strength, and respiratory parameters will be evaluated at baseline and study completion.

The findings will provide objective data on the effectiveness of WBV and NMES in ICU patients, guiding future research and treatment while contributing to national and international literature.

DETAILED DESCRIPTION:
This randomized controlled trial will investigate and compare the effects of WBV and NMES on respiratory muscle strength, respiratory parameters, and muscle mass, composition, elasticity, and strength in ICU patients. A total of 45 patients will be randomly assigned to one of three groups:

WBV Group (n=15): Conventional therapy + Whole Body Vibration NMES Group (n=15): Conventional therapy + Neuromuscular Electrical Stimulation Control Group (n=15): Conventional therapy only

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years,
* Clinically stable condition,
* Deemed suitable for physiotherapy interventions by the intensive care specialist physician,
* Willing to participate in the study or, if unconscious, authorized by a first-degree relative.

Exclusion Criteria:

* Patients with coagulation disorders (Prothrombin Time (PT); International Normalized Ratio (INR) value greater than 1.5, and platelet count less than 50,000/mm³),
* Agitated patients (Richmond Agitation and Sedation Scale (RASS) score ≥ 2)
* Patients with signs of increased intracranial pressure,
* Patients with cardiac and respiratory instability (respiratory rate above 30 breaths/min, systolic blood pressure below 80 mmHg or above 200 mmHg, diastolic blood pressure below 50 mmHg or above 100 mmHg, PaO₂ < 65 mmHg, FiO₂ > 55%),
* Patients with hemodynamic instability (requiring dopamine support > 5 mcg/kg/min),
* Patients in shock,
* Patients with malignancies,
* Pregnant individuals,
* Patients using pacemakers,
* Patients with high fever.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of Muscle Thickness | at 4 weeks
  The patient's muscle thickness is evaluated with the EDAN DUS 60 ultrasonography device, and the increase in muscle thickness is measured.
Muscle Elasticity Assessment | 4 weeks
  Myoton device will be used for the assessment. How the values change according to the application will be examined.
Muscle Strength Assessment | 4 weeks
  Muscle strength will be objectively measured using a myometer in conjunction with the Medical Research Council (MRC) scale. Each muscle group is assessed on a scale from 0 (no movement or complete paralysis) to 5 (full normal strength). The cumulative MRC scale score ranges from 0 to 60, with a score below 48 indicating the presence of muscle weakness.
Grip Strength Assessment | 4 weeks
  Grip strength will be measured using a Jamar brand dynamometer. Hand grip strength provides information about overall body muscle strength.
Measurement of Respiratory Muscle Strength | 4 weeks
  To measure respiratory muscle strength, patients connected to mechanical ventilation will be switched to the CPAP mode of the ventilator. The ventilator settings will be adjusted to PEEP: 5 cmH2O and Psup: 10 cmH2O to overcome the physiological resistance of the ventilator circuit. The pressure value displayed on the mechanical ventilator screen will be recorded as the MIB value
Functional Status Assessment | 4 weeks
  The Premorbid Activity Level Scale will be used to determine the patient's functional status in daily life prior to intensive care. This scale categorizes activity levels from 0 (completely dependent) to 4 (independent in all activities). . The P-FIT is scored from 0 to 12, with higher scores indicating better physical function.
Functional Status Assessment | 4 weeks
  The CPAX is scored from 0 to 50, where higher scores reflect greater independence and physical ability.
Assessment of Inspiratory tidal volume | 4 weeks
  Inspiratory tidal volume (TVi) in milliliters in L/min will be recorded.
Assessment of Expiratory tidal volume | 4 weeks
  Expiratory tidal volume (TVe) in milliliters in L/min will be recorded.
Assessment of Minute Ventilation | 4 weeks
  Minute ventilation in L/min will be recorded.

SECONDARY OUTCOMES:
Assessment of APCAHE II | 4 weeks
  APACHE II ranges from 0 to 71, combining physiological, laboratory, and demographic data to predict severity and mortality risk.The higher the APACHE II score, the higher the patient's risk of mortality in the intensive care unit.
Consciousness Level Assessment | 4 weeks
  The Glasgow Coma Scale (GCS) will be used to determine the patient's level of consciousness. The Glasgow Coma Scale (GCS) assesses consciousness by evaluating three components: eye opening (4-1), verbal response (5-1), and motor response (6-1). Scores range from 3 (deep coma) to 15 (fully alert), with lower scores indicating more severe impairment. A score of 8 or below typically suggests the need for immediate intervention.
Agitation, Anxiety, and Sedation Assessment | 4 weeks
  Agitation and anxiety levels will be assessed using the Richmond Agitation and Sedation Scale (RASS).. Scores range from +4 (combative) to 0 (calm and alert) to -5 (unarousable). Positive scores indicate agitation, 0 indicates normal alertness, and negative scores reflect increasing levels of sedation.
Pain Assessment-The Nonverbal Pain Scale | 4 weeks
  The Nonverbal Pain Scale (NVPS) is designed for adults who cannot communicate verbally and evaluates pain based on five categories: facial expression, body movement, muscle tension, compliance with ventilation, and vocalization, each scored from 0 to 2, with a total score ranging from 0 to 10. A score closer to 10 suggests severe pain, while a score closer to 0 indicates minimal or no pain.
Dyspnea Assessment | 4 weeks
  Patients will rate their dyspnea by marking a point on a 10 cm horizontal line, where 0 represents no fatigue and 10 indicates the worst fatigue imaginable. The score is determined by measuring the distance from the 0 point to the patient's mark, providing a quantitative measure of dyspnea intensity.
SOFA Assessment | 4 weeks
  SOFA evaluates dysfunction in six organ systems, with a total score ranging from 0 to 24, where higher scores indicate greater dysfunction and mortality risk
Pain Assessment-The Visual Analog Scale | 4 weeks
  The Visual Analog Scale (VAS) is a self-reported measure where patients mark their pain intensity on a 10 cm line, with 0 indicating no pain and 10 representing the worst pain imaginable.
General Body Fatigue Assessment | 4 weeks
  Patients will rate their fatigue by marking a point on a 10 cm horizontal line, where 0 represents no fatigue and 10 indicates the worst fatigue imaginable. The score is determined by measuring the distance from the 0 point to the patient's mark, providing a quantitative measure of fatigue intensity.
Heart Rate Assessment | at 4 weeks
  The heart rate will be recorded on the monitor at the beginning, end and half an hour after the session.
Systolic Pressure Assessment | at 4 weeks
  Systolic pressure will be recorded on the monitor at the beginning, end and half an hour after the session.
Diastolic Pressure Assessment | at 4 weeks
  Diastolic Pressure will be recorded on the monitor at the beginning, end and half an hour after the session.
Oxygen Saturation Assessment | at 4 weeks
  Oxygen saturation will be recorded on the monitor at the beginning, end and half an hour after the session.
Respiratory Rate Assessment | at 4 weeks
  The respiratory rate will be recorded at the beginning, end and half an hour after the session.

CONTACTS AND LOCATIONS:
Locations (1):
- Istınye University, Istanbul, Turkey (Türkiye)